CLINICAL TRIAL: NCT03617731
Title: A Randomized Phase III Trial Assessing the Benefit of the Addition of Isatuximab to Lenalidomide / Bortezomib / Dexamethasone (RVd) Induction and Lenalidomide Maintenance in Patients With Newly Diagnosed Multiple Myeloma
Brief Title: Trial on the Effect of Isatuximab to Lenalidomide/Bortezomib/Dexamethasone (RVd) Induction and Lenalidomide Maintenance in Patients With Newly Diagnosed Myeloma (GMMG HD7)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Heidelberg Medical Center (Other)
Responsible Party: Principal Investigator, Prof. Dr. Hartmut Goldschmidt, Head of Division of Multiple Myeloma, University of Heidelberg Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GMMG HD7
Record Dates: First submitted 2018-07-24; First posted 2018-08-06 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; Bortezomib; Dexamethasone; isatuximab

STUDY DESIGN:
Intervention Model Description: 2 x 2 arms, 1. randomization before induction therapy (arm IA and IB), 2. randomization before maintenance therapy (arm IIA and IIB)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- IA (Active Comparator): Patients in arm IA are treated with 3 cycles RVd (lenalidomide 25 mg/d p.o. d1 - 14 and d22 - 35; bortezomib 1.3 mg/m2 s.c. d1, 4, 8, 11, 22, 25, 29, 32; dexamethasone p.o. 20 mg/d d1-2, 4-5, 8-9, 11-12, 15, 22-23, 25-26, 29-30, 32-33).Treatment repeats every 42 days (d43 = cycle 2 d1). Standard intensification: For all patients, stem cells are mobilized by GMMG Standard protocols (CAD: cyclophosphamide, doxorubicin, dexamethasone) and G-CSF. At least 7.5x106 CD34+ cells/kg body weight are harvested. High dose treatment (melphalan 200mg/m², HDT) followed by autologous stem cell transplantation (ASCT) is started 4 - 6 weeks after CAD. For patients not in CR after HDT1, a second HDT is performed within 3 months.
  Interventions: Drug: Lenalidomide; Drug: Bortezomib; Drug: Dexamethasone
- IB (Experimental): Patients in arm IB are treated with 3 cycles RVd + Isatuximab (lenalidomide 25 mg/d p.o. d1 - 14 and d22 - 35; bortezomib 1.3 mg/m2 s.c. d1, 4, 8, 11, 22, 25, 29, 32;dexamethasone p.o. 20 mg/d d1-2, 4-5, 8-9, 11-12, 15, 22-23, 25-26, 29-30, 32-33).Isatuximab (10 mg/kg i.v. C1: d 1, 8, 15, 22, 29; C2-3: d 1, 15, 29).Treatment repeats every 42 days (d43 = cycle 2 d1). Standard intensification: For all patients, stem cells are mobilized by GMMG Standard protocols (CAD: cyclophosphamide, doxorubicin, dexamethasone) and G-CSF. At least 7.5x106 CD34+ cells/kg body weight are harvested. High dose treatment (melphalan 200mg/m², HDT) followed by autologous stem cell transplantation (ASCT) is started 4 - 6 weeks after CAD. For patients not in CR after HDT1, a second HDT is performed within 3 months.
  Interventions: Drug: Lenalidomide; Drug: Bortezomib; Drug: Dexamethasone; Drug: Isatuximab
- IIA (Active Comparator): maintenance treatment with Lenalidomide 10mg/d (increased to 15mg/d after 3 months) repeated every 28d. Maintenance treatment is planned for up to 36 months or until progression if progression occurs first.
  Interventions: Drug: Lenalidomide
- IIB (Experimental): maintenance treatment with Lenalidomide 10mg/d (increased to 15mg/d after 3 months) + Isatuximab (10 mg/kg; C1: d1, 8, 15, 22; C2-C3: d1 + 15; C4-39:d1, repeated every 28d). Within the trial, maintenance treatment is planned for up to 36 months or until progression if progression occurs first.
  Interventions: Drug: Lenalidomide; Drug: Isatuximab

INTERVENTIONS:
Drug: Lenalidomide — 25 mg per os on day 1-14 and d22-35 in induction cycle 1-3 (Arms IA and IB) 10 mg p.o. on day 1-28 in maintenance cycle 1-3, 15 mg p.o. on day 1-28 in maintenance cycle 4-39 (Arms IIA and IIB)
  Other Names: Revlimid
Drug: Bortezomib — all arms: 1,3 mg/m^2 subcutaneous on day 1, 4, 8, 11, 22, 25, 29 32 in 3 induction cycles
  Other Names: Velcade
  Arms: IA; IB
Drug: Dexamethasone — 20 mg per os on day 1,2 and 4,5 and 8,9 and 11,12 and 15 and 22,23 and 25,26 and 29,30 and 32,33 in induction cycles 1-3 (Arms IA and IB). Maintenance cycle 1 on day 1, 8, 15, 22 Dexamethasone 20 mg/d per os (Arm IIA). In Arm IIB Dexamethasone 20 mg i.v. on days of Isatuximab infusion in the first maintenance cycle (d 1, 8, 15, 22), dexamethasone will be administered intravenously as part of the premedication. If an isatuximab dose is skipped or discontinued dexamethasone should be administered orally.
  Arms: IA; IB
Drug: Isatuximab — 10 mg/kg in the vein( i.v) on day 1,8,15, 22, 29 in induction cycle 1 on day 1, 15 and 29 in induction cycle 2 and 3 (Arm IB). 10 mg/kg i.v. on day 1,8, 15 and 22 in maintenance cycle 1, 10 mg/kg i.v. on day 1 and 15 in maintenance cycle 2 and 3, 10 mg/kg i.v. on day 1 in maintenance cycle 4 - 39 (Arm IIB)
  Arms: IB; IIB

SUMMARY:
Trial in patients with newly diagnosed myeloma to evaluate the effect of isatuximab in induction therapy with lenalidomide/bortezomib/dexamethasone (RVd) and in lenalidomide maintenance treatment

DETAILED DESCRIPTION:
Prospective, multicentre, randomised, parallel group, open, phase III clinical trial, for patients with confirmed diagnosis of untreated multiple myeloma requiring systemic therapy.

Investigational Medicinal Products: Isatuximab, Lenalidomide

1. Randomization: Patients are randomized in one of 2 study arms (IA or IB) before induction therapy. Patients randomized in arm IA will receive 3 cycles RVd (Bortezomib (Velcade®), Lenalidomide (Revlimid®, each cycle is 42 days), Dexamethasone). Patients in arm IB will additionally receive the monoclonal antibody Isatuximab in the 3 cycles RVd. After induction therapy patients undergo intensifying therapy according to GMMG standard (usually mobilization therapy followed by stem cell collection and autologous stem cell transplantation).
2. Randomization: Before maintenance treatment patients are randomized in one of 2 study arms (IIA and IIB): Patients in arm IIA receive Lenalidomide maintenance therapy for three years, patients in arm IIB receive additional Isatuximab.

There are two primary objectives:

1. to compare the induction regimen (IA vs IB) regarding minimal residual disease (MRD) negativity after induction (assessed by flow cytometry; sensitivity at least 1e-5)
2. to compare the maintenance strategies (arms IIA vs IIB) regarding progression-free survival (PFS), defined as time from 2nd randomization (prior to maintenance therapy) to progression or death from any cause whichever occurs first.

The duration of the trial for each patients is expected to be 45-48 months (induction and intensification treatment: 6-9 months, 3 months rest between intensification and start of maintenance phase 36 months).

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of untreated multiple myeloma requiring systemic therapy (diagnostic criteria (IMWG updated criteria (2014)1) see appendix IA. For some patients systemic therapy may be required though these diagnostic criteria are not fulfilled. In this case the GMMG study office has to be consulted prior to inclusion.)
2. Patient is eligible for high dose therapy and autologous stem cell transplantation.
3. Measurable disease, defined as any quantifiable monoclonal protein value, defined by at least one of the following three measurements:2

   * Serum M-protein ≥ 10g/l (for IgA ≥ 5g/l)
   * Urine light-chain (M-protein) of ≥ 200 mg/24 hours
   * Serum FLC assay: involved FLC level ≥ 10 mg/dl provided sFLC ratio is abnormal
4. Age 18 - 70 years inclusive
5. WHO performance status 0-2
6. Negative pregnancy test at inclusion (females of childbearing potential)
7. All patients must agree on the requirements regarding the lenalidomide pregnancy prevention plan described in section 6. For all men and females of childbearing potential: patients must be willing and capable to use adequate contraception during the complete therapy.
8. All patients must

   * agree to abstain from donating blood while taking lenalidomide and for 28 days following discontinuation of lenalidomide therapy
   * agree not to share study drug lenalidomide with another person and to return all unused study drug to the investigator or pharmacist
9. Ability of patient to understand character and individual consequences of the clinical trial
10. Provide written informed consent (must be available before enrolment in the trial)

Exclusion Criteria

1. Patient has known hypersensitivity (or contraindication) to dexamethasone, sucrose histidine (as base and hydrochloride salt), boron, mannitol, and polysorbate 80 or any of the components of study therapy that are not amenable to premedication with steroids or H2 blockers that would prohibit further treatment with these agents.
2. Systemic AL amyloidosis (except for AL amyloidosis of the skin or the bone marrow)
3. Plasma cell leukemia
4. Previous chemotherapy or radiotherapy during the past 5 years except local radiotherapy in case of local myeloma progression. (Note: patients may have received a cumulative dose of up to 160 mg of dexamethasone or equivalent as emergency therapy.) Previous therapy due to smouldering myeloma may be acceptable. In this case the GMMG study office has to be consulted prior to inclusion
5. Severe cardiac dysfunction (NYHA classification III-IV), ejection fraction < 40%
6. Significant hepatic dysfunction (ASAT and/or ALAT ≥ 3 times normal level and/or serum bilirubin ≥ 1.5 times normal level if not due to hereditary abnormalities as Gilbert's disease), unless related to myeloma.
7. Patients with active or history of hepatitis B or C
8. HIV positivity
9. Patients with active, uncontrolled infections
10. Patients with severe renal insufficiency (Creatinine Clearance < 30ml/min)
11. Patients with peripheral neuropathy or neuropathic pain, CTC grade 2 or higher (as defined by the NCI Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.0)
12. Patients with a history of active malignancy during the past 5 years with the exception of following malignancies after curative therapy: basal cell carcinoma of the skin, squamous cell skin carcinoma, stage 0 cervical carcinoma or any in situ malignancy
13. Patients with acute diffuse infiltrative pulmonary and/or pericardial disease
14. Autoimmune hemolytic anemia with positive Coombs test or immune thrombocytopenia
15. Platelet count < 75 x 109/l
16. Haemoglobin < 8.0 g/dl, unless related to myeloma
17. Absolute neutrophil count (ANC) < 1.0 x 109/l (the use of colony stimulating factors within 14 days before the test is not allowed)
18. Corrected serum calcium > 14 mg/dl (> 3.5 mmol/l)
19. Unable or unwilling to undergo thromboprophylaxis
20. Pregnancy and lactation
21. Participation in other clinical trials. This does not include long-term follow-up periods without active drug treatment of previous studies during the last 6 months.
22. Prisoners or subjects who are legally institutionalized, or those unwilling or unable to comply with scheduled visits, drug administration plan, laboratory tests, other study procedures, and study restrictions.

No patients will be allowed to enrol in this trial more than once.

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 662 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
MRD negativity after induction Treatment (comparison of arms IA and IB) | 18 weeks after start of study treatment
  Detection of minimal residual disease by flow cytometry (sensitivity at least 1e-5)
Progression Free Survival (PFS) after second randomization (arms IIA and IIB) | time from 2. randomization to progression or death from any cause whichever comes first, censored after three years of maintenance therapy
  Response Evaluation by IMWG criteria

SECONDARY OUTCOMES:
to compare the four treatment arms (IA-IIA, IA-IIB, IB-IIA, IB-IIB) regarding Progression free survival (PFS) | time from 1. randomization (study inclusion) to progression or death whichever comes first (assessed up to 79 months)
  Response evaluation by IMWG criteria
to compare all 4 treatment arms (IA-IIA, IA-IIB, IB-IIA, IB-IIB) regarding overall survival (OS) from time of 1.randomization | time from randomisation to time of death from any cause (assessed up to 79 months)
  survival status
Overall survival from second randomization | time from 2. randomization to time of death from any cause (assessed up to 75 months)
  survival status
Complete Response (CR) rates after induction therapy | After induction treatment (18 weeks after start of treatment)
  Response Evaluation by IMWG criteria
Complete Response (CR) after high dose therapy | After high dose therapy (9 or 12 months after start of therapy)
  Response Evaluation by IMWG criteria
Complete Response (CR) during/after maintenance therapy | During/after maintenance therapy (6 months after start of therapy up to 36 months of maintenance therapy)
  Response Evaluation by IMWG criteria
MRD negativity after high dose therapy | After high dose therapy (9 or 12 months after start of therapy)
  Detection of minimal residual disease by flow cytometry (sensitivity at least 1e-5)
MRD negativity during and after maintenance therapy | up to 36 months after start of maintenance therapy
  Detection of minimal residual disease by flow cytometry (sensitivity at least 1e-5)
Best response to treatment during the trial | response assessment after 3 months, 4,5 months, 5,5 months, 9 months (if applicable: 3 months later after 2. high dose therapy) subsequently every 3 months during maintenance treatment, up to 48 months after start of study treatment
  Response evaluation by IMWG criteria
PFS 2 (PFS after next line of therapy) from 2. randomization | time from 2. randomization to time of overall end of trial (up to 75 months)
  Response evaluation by IMWG criteria
Toxicity during induction and maintenance with respect to adverse events of CTC grade >3 (and specific adverse events of CTC grade > 2 as defined in the protocol and serious adverse events | : from first administration of study drug until 30 days after last administration of study drug or any drug of the study treatment or upon start of a new subsequent chemotherapy, whichever occurs first
  toxicity according CTCAE Version v5.0
Quality of Life Assessment | assessed at baseline, after ca. 4.5 months, 9 months, (additionally after 12 months,if a second high dose therapy is administered) after 12 months of maintenance and at end of study (up to 50 months)
  EORTC (European Organization of Research and Treatment of Cancer) -QLQC30 Questionnaire to assess the quality of life of cancer patients. Impairment of daily life is asked in 4 scales from "not at all" (best) to "very much" (worst scale), EORTC-QLQMY20 questionnaire to assess health-related quality of life in patients with multiple myeloma with 4 scales from "not at all (best scale) to "very much" (worst scale); EQ(EuroQol Group)-5D-5L Health questionnaire comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. Additionally a visual analogue scale from 100 (best) to 0 (worst scale) is used to assess the quality of health questionnaires.
Pharmakokinetic analyses of Isatuximab in induction treatment of patients in Arm IB (selected sites only) | Up to 18 weeks in induction treatment (C1: D1, before infusion, at end of infusion, 1 h after infusion, C1 D8,15,22,29 before infusion; C2 and 3:D1 before infusion
  Determination of serum concentration of isatuximab at different timepoints before, during and after isatuximab infusion
Pharmakokinetic analyses of Isatuximab in maintenance treatment of patients in Arm IIB (selected sites only) | Up to 9 months (C1: D1, before infusion, at end of infusion, 1 h after infusion, C1 D8,15,22 before infusion, C2 -9, D1: before infusion
  Determination of serum concentration of isatuximab at different timepoints

CONTACTS AND LOCATIONS:
Overall Officials: Hartmut Goldschmidt, Prof. Dr., Principal Investigator — Med. Klinik V, University Hospital Heidelberg
Locations (72):
- Germany (72):
  - Uniklinik RWTH Aachen, Klinik für Hämatologie, Onkologie, Hämostaseologie und Stammzelltransplantation, Aachen
  - Helios Klinikum Bad Saarow, Klinik für Hämatologie, Onkologie und Palliativmedizin, Bad Saarow
  - Charité, Campus Benjamin Franklin , III. Medizinische Abteilung (Hämatologie/Onkologie), Berlin
  - Vivantes Klinikum Neukölln, Klinik für Hämatologie und Onkologie, Berlin
  - HELIOS Klinikum, Klinik für Hämatologie, Onkologie und Immunologie, Berlin
  - Studiengesellschaft Onkologie Bielefeld GbR, Bielefeld
  - Klinikum Bielefeld, Klinik für Hämatologie, Onkologie und Palliativmedizin, Bielefeld
  - Medizinische Universitätsklinik, Knappschaftskrankenhaus, Bochum
  - Universitätsklinikum Bonn, Medizinische Klinik und Poliklinik III, Schwerpunkt Onkologie, Hämatologie und Rheumatologie, Bonn
  - Johanniter Krankenhaus Bonn, Bonn
  - Zentrum für ambulante Hämatologie und Onkologie (ZAHO), Bonn
  - Städtisches Klinikum Braunschweig, Med. Klinik III, Hämatologie und Onkologie, Braunschweig
  - Klinikum Chemnitz GmbH, Innere Medizin III, Chemnitz
  - Uniklinik Köln, Klinik I für Innere Medizin, Cologne
  - Carl-Thiem-Klinikum Cottbus gGmbH, II. Medizinische Klinik, Cottbus
  - Onkologisches Studienzentrum Darmstadt, Darmstadt
  - Klinikum Darmstadt, Med. Klinik V, Hämatologie/Onkologie, Darmstadt
  - Universitätsklinikum Carl Gustav Carus Dresden, an der Technischen Universität Dresden, Medizinische Klinik und Poliklinik I, Dresden
  - HELIOS St. Johannes Klinik, Akademisches Krankenhaus der Heinrich-Heine-Universität Düsseldorf, Duisburg
  - Marien Hospital Düsseldorf GmbH, Klinik für Onkologie, Hämatologie und Palliativmedizin, Düsseldorf
  - Universitätsklinikum Düsseldorf, Klinik für Hämatologie,Onkologie und Klin. Immunologie, Düsseldorf
  - Universitätsklinik Erlangen, Erlangen
  - St. Antonius-Hospital Eschweiler, Klinik für Hämatologie / Onkologie, Eschweiler
  - Universitätsklinikum Essen, Klinik für Hämatologie, Essen
  - Ev. Krankenhaus Essen-Werden gGmbH, Zentrum für Innere Medizin, Klinik für Hämatologie, Onkologie und Stammzelltransplantation, Essen
  - Gemeinschaftspraxis Prof. Dr. Michael Kiehl und Dipl. Med. Wolfgang Stein, Frankfurt (Oder)
  - Klinikum Frankfurt (Oder) GmbH, Frankfurt (Oder)
  - Centrum für Hämatologie und Onkologie Bethanien, Frankfurt am Main
  - Agaplesion Markus Krankenhaus, Med. Klinik I, Frankfurt am Main
  - Krankenhaus Nordwest, Institut für Klinisch-Onkologische Forschung, Frankfurt am Main
  - Universitätsklinikum Frankfurt, Goethe-Universität Medizinische Klinik II, Frankfurt am Main
  - Klinikum Fulda, Klinisches Studienzentrum GmbH, Fulda
  - Universitätsklinik der Justus-Liebig-Universität, Medizinische Klinik IV, Giessen
  - Katholisches Karl-Leisner-Klinikum gGmbH, Wilhelm-Anton-Hospital Goch, Klinik für Hämatologie - Onkologie, Goch
  - Kath. Krankenhaus Hagen gGmbH, Abt. Hämatologie/Onkologie, Hagen
  - Asklepios Klinik Hamburg St. Georg, Hamburg
  - Universitätsklinikum Hamburg Eppendorf, Zentrum für Onkologie, Studienzentrale der II. Medizinischen Klinik, Hamburg
  - Asklepios Klinik Hamburg Altona, II. Med. Klinik, Hamburg
  - Immunologisch-onkologisches MVZ am Siloah Krankenhaus, Hanover
  - KRH Klinikum Siloah, Klinik für Hämatologie und Onkologie, Hanover
  - Onkologische Schwerpunktpraxis Heidelberg, Heidelberg
  - Krankenhaus St. Vincentius der evangelischen Stadtmission Heidelberg, Abt. Hämatologie, Onkologie, Rheumatologie, Heidelberg
  - University Hospital Heidelberg, Med. Klinik V, Heidelberg
  - SLK Kliniken Heilbronn, Med. Klinik III, Heilbronn
  - Marien Hospital Herne, Herne
  - Universitätsklinikum des Saarlandes, Innere Medizin I, Homburg (Saar)
  - Westpfalz-Klinikum GmbH, Klinik für Innere Medizin I, Kaiserslautern
  - Städtisches Klinikum Karlsruhe, Karlsruhe
  - Praxisklinik für Hämatologie und Onkologie, Koblenz
  - Gemeinschaftspraxis für Hämatologie und Onkologie am Caritas Krankenhaus, Lebach
  - Universitätsklinikum Leipzig AöR, Medizinische Klinik und Poliklinik I-Hämatologie und Zelltherapie, Internistische Onkologie, Hämostaseologie, Leipzig
  - Med. Klinik A, Klinikum der Stadt Ludwigshafen am Rhein gGmbH, Ludwigshafen am Rhein
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, III. Med. Klinik, Mainz
  - III. Medizinische Klinik Hämatologie und Internistische Onkologie, Mannheim
  - Mannheimer Onkologie Praxis, Mannheim
  - Philipps-Universität Marburg, Hämatologie/Onkologie/Immunologie, Marburg
  - Mühlenkreiskliniken (AöR) Johannes Wesling Klinikum Minden, Hämatologie/Onkologie, Hämostaseologie und Palliativmedizin, Minden
  - Krankenhaus Maria Hilf GmbH, Franziskuskrankenhaus, Med. Klinik I, Mönchengladbach
  - Universitätsklinikum Münster, Med. Klinik A, Münster
  - Klinikum Osnabrück GmbH, Osnabrück
  - Brüderkrankenhaus St. Josef Paderborn, Klinik für Hämatologie und Onkologie, Paderborn
  - Krankenhaus Barmherzige Brüder, Klinik für Onkologie und Hämatologie, Regensburg
  - Gemeinschaftspraxis für Hämatologie und Onkologie, Onkologisches Zentrum, Saarlouis
  - Diakonie-Klinikum Schwäbisch Hall gGmbH, Innere Medizin III, Schwäbisch Hall
  - ZAHO-Zentrum für ambulante Hämatologie und Onkologie, Standort Siegburg, Siegburg
  - Onkologische Schwerpunktpraxis Speyer, Speyer
  - Klinikum Stuttgart, Stuttgart Cancer Center, Tumorzentrum Eva Mayr-Stihl, Stuttgart
  - Klinikum Mutterhaus der Borromäerinnen gGmbH, Trier
  - University Hospital Tübingen, Med. Klinik und Poliklinik, Abt. II, Tübingen
  - Bundeswehrkrankenhaus Ulm, Abteilung Innere Medizin - Hämatologie und internistische Onkologie, Ulm
  - Schwarzwald-Baar Klinikum, Innere Medizin II, Villingen-Schwenningen
  - Rems-Murr-Kliniken gGmbH, Winnenden

REFERENCES:
- [Derived] Mai EK, Bertsch U, Pozek E, Fenk R, Besemer B, Hanoun C, Schroers R, von Metzler I, Hanel M, Mann C, Leypoldt LB, Heilmeier B, Huhn S, Vogel SK, Hundemer M, Scheid C, Blau IW, Luntz S, Weinhold N, Tichy D, Holderried TAW, Trautmann-Grill K, Gezer D, Klaiber-Hakimi M, Muller M, Shumilov E, Knauf W, Michel CS, Geer T, Riesenberg H, Lutz C, Raab MS, Benner A, Hoffmann M, Weisel KC, Salwender HJ, Goldschmidt H; German-Speaking Myeloma Multicenter Group (GMMG) HD7 Investigators; German-speaking Myeloma Multicenter Group (GMMG) HD7. Isatuximab, Lenalidomide, Bortezomib, and Dexamethasone Induction Therapy for Transplant-Eligible Newly Diagnosed Multiple Myeloma: Final Part 1 Analysis of the GMMG-HD7 Trial. J Clin Oncol. 2025 Apr 10;43(11):1279-1288. doi: 10.1200/JCO-24-02266. Epub 2024 Dec 9. PMID 39652594
- [Derived] Mai EK, Hielscher T, Bertsch U, Salwender HJ, Zweegman S, Raab MS, Munder M, Pantani L, Mancuso K, Brossart P, Beksac M, Blau IW, Durig J, Besemer B, Fenk R, Reimer P, van der Holt B, Hanel M, von Metzler I, Graeven U, Muller-Tidow C, Boccadoro M, Scheid C, Dimopoulos MA, Hillengass J, Weisel KC, Cavo M, Sonneveld P, Goldschmidt H. Predictors of early morbidity and mortality in newly diagnosed multiple myeloma: data from five randomized, controlled, phase III trials in 3700 patients. Leukemia. 2024 Mar;38(3):640-647. doi: 10.1038/s41375-023-02105-6. Epub 2023 Dec 7. PMID 38062124
- [Derived] Kauer J, Freundt EP, Schmitt A, Weinhold N, Mai EK, Muller-Tidow C, Goldschmidt H, Raab MS, Kriegsmann K, Sauer S. Stem cell collection after lenalidomide, bortezomib and dexamethasone plus elotuzumab or isatuximab in newly diagnosed multiple myeloma patients: a single centre experience from the GMMG-HD6 and -HD7 trials. BMC Cancer. 2023 Nov 21;23(1):1132. doi: 10.1186/s12885-023-11507-9. PMID 37990162
- [Derived] Goldschmidt H, Mai EK, Bertsch U, Fenk R, Nievergall E, Tichy D, Besemer B, Durig J, Schroers R, von Metzler I, Hanel M, Mann C, Asemissen AM, Heilmeier B, Weinhold N, Huhn S, Kriegsmann K, Luntz SP, Holderried TAW, Trautmann-Grill K, Gezer D, Klaiber-Hakimi M, Muller M, Khandanpour C, Knauf W, Scheid C, Munder M, Geer T, Riesenberg H, Thomalla J, Hoffmann M, Raab MS, Salwender HJ, Weisel KC; German-Speaking Myeloma Multicenter Group (GMMG) HD7 investigators. Addition of isatuximab to lenalidomide, bortezomib, and dexamethasone as induction therapy for newly diagnosed, transplantation-eligible patients with multiple myeloma (GMMG-HD7): part 1 of an open-label, multicentre, randomised, active-controlled, phase 3 trial. Lancet Haematol. 2022 Nov;9(11):e810-e821. doi: 10.1016/S2352-3026(22)00263-0. PMID 36328040